CLINICAL TRIAL: NCT06829264
Title: A Pilot Trial of the Individualized Placement and Support Model in Autistic Adults in the Community
Brief Title: Testing an Evidence-Based Supported Employment Model in Autistic Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024578
Record Dates: First submitted 2025-01-24; First posted 2025-02-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group - Agencies Receiving IPS (Experimental): Participating agencies will be randomized, with 2/3 of agencies receiving IPS first. The estimated total number of agencies = 6 (each referring 10 consumers), meaning that 4 agencies (40 clients) would be assigned to receive IPS training first. These agencies will be expected to deliver IPS services for a duration of 12 months.
  Interventions: Behavioral: Individualized Placement and Support Model
- Control Group - Agencies Receiving Supportive Employment Intervention (Active Comparator): One third of the agencies (approximately 2 agencies and 20 consumers) will be assigned to the wait-list control group will continue to provide their usual services during the first 12 months. In addition, clients of these agencies will be offered a Supportive Employment Intervention, which includes weekly sessions offering support with some help on employment-related skills such as resume building, job interviewing, and workplace communication strategies.
  Interventions: Behavioral: Supportive Employment Intervention

INTERVENTIONS:
Behavioral: Individualized Placement and Support Model — The Individualized Placement and Support (IPS) model is an evidence-based approach to supported employment designed to help individuals with disabilities achieve and maintain competitive integrated employment (CIE). IPS emphasizes person-centered planning, rapid engagement, and focusing on individual strengths and preferences. Key features include prioritizing CIE, eligibility based on the desire to work, integration of employment services with mental health support, rapid job searches, tailored job development, and time-unlimited, individualized support. IPS also provides benefits counseling to help participants manage employment while maintaining government benefits. For this study, IPS is adapted to meet the needs of autistic individuals by enhancing provider training and family involvement to improve outcomes.
  Arms: Treatment Group - Agencies Receiving IPS
Behavioral: Supportive Employment Intervention — This intervention consists of a weekly series of sessions designed for adult consumers, incorporating supportive elements inspired by the ACCESS (Acquiring Career, Coping, Executive, and Social Skills) program developed at the UC Davis MIND Institute. The sessions will provide time to discuss consumer experiences, give general guidance and some training in employment-related skills, including resume building, job interviewing, and strategies for giving and receiving feedback in the workplace.
  Arms: Control Group - Agencies Receiving Supportive Employment Intervention

SUMMARY:
This study aims to enhance employment outcomes for young adults with autism and intellectual and developmental disabilities (IDD) through the implementation of an evidence-based supported employment model known as Individual Placement and Support for Autism (IPS-AUT). The study will evaluate the feasibility, acceptability, and effectiveness of IPS-AUT in promoting Competitive Integrated Employment (CIE). The trial will involve partnerships with supported employment agencies, training providers in IPS-AUT, and assessing employment outcomes and implementation factors. The ultimate goal is to create a scalable, evidence-based employment support model for individuals with autism.

DETAILED DESCRIPTION:
This study builds on prior research and pilot testing of IPS in the autism and IDD community by implementing a 12-month Hybrid Type 1 trial to evaluate the effectiveness and implementation of IPS-AUT. The current study will include three primary aims:

Consumer Support Toolbox Development: Using data from previous focus groups, researchers will develop and test a Consumer Support Toolbox (CST) to align IPS services with autistic consumer needs.

IPS-AUT Implementation and Outcomes Evaluation: A 12-month Hybrid Type 1 trial will assess feasibility, acceptability, fidelity to IPS standards, and employment outcomes. The study aims for a minimum 50% success rate in Competitive Integrated Employment and at least 75% feasibility and acceptability.

Mediators of Employment Outcomes: Researchers will explore the role of parent/carer engagement and work-related social cognition in improving employment success.

This trial is designed to prepare for a larger R01-funded study by refining implementation strategies and addressing key barriers. Participants will include young adults with autism, their employment providers, and caregivers, with data collected through surveys, focus groups, interviews, and standardized assessments. The study is funded by the National Institute of Mental Health and conducted in collaboration with supported employment agencies in California.

ELIGIBILITY:
Inclusion Criteria: California supported employment agency clients meeting the following criteria:

* Community diagnosis of autism spectrum disorder, demonstrated by a letter from a healthcare provider, psychologist, other mental health professional, Regional Center representative, or school psychologist.
* Aged 18-40 years.
* Minimum 4th-grade reading level (approximately mild ID).
* Not currently employed but seeking employment.

Exclusion Criteria:

- Not interested in employment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of IPS Implementation | 18 months
  Measure: Agency feasibility ratings and IPS fidelity reviews. Assessment Method: Trained IPS fidelity reviews will assess fidelity using the IPS Fidelity Scale (Bond et al., 2012) at baseline, 6 months, and 12 months. Additionally, feasibility will be assessed through participant, parent, and provider ratings on a 5-point Likert scale (1 = not feasible at all, 5 = highly feasible).
  Expect outcome: Achieve good fidelity at the 12-month fidelity review. Achieve at least 75% feasibility.
Competitive Integrated Employment (CIE) Attainment | 18 months
  Measure: CIE attainment log Assessment Method: Monthly reports on employment status will be collected via phone or in virtual meetings with providers. Employment status will be categorized as "Employed in CIE," "Not Employed," or "Transitioned Out of CIE." Expect outcome: Minimum of 50% CIE attainment success.
Competitive Integrated Employment (CIE) Retention | 18 months
  Measure: CIE retention log Assessment Method: Monthly reports on employment status will be collected via phone or in virtual meetings with providers. Employment status will be verified as "Employed in CIE," "Not Employed," or "Transitioned Out of CIE." Expect outcome: Minimum of 50% CIE retention.
Acceptability of IPS Implementation | 18 months
  Measure: Participant, parent, and provider satisfaction. Assessment Method: Surveys using a 5-point Likert scale (1 = not satisfied at all, 5 = very satisfied) to assess satisfaction with IPS services and overall perceived value of the intervention.
  Expect outcome: Achieve at least 75% acceptability.
Parent/Carer Engagement | 18 months
  Measure: Family Engagement Survey Assessment Method: Monthly surveys will be collected via phone or online to collect information on family involvement and satisfaction with the services their family member is receiving. Family members/carers will rate their involvement and satisfaction on a Likert scale survey.
Work-Related Social Cognition | 18 months
  Work-related social cognition is evaluated to understand its impact on functional outcomes such as planning, problem-solving, and attention, which are critical to employment success.
  Assessment Method: The Adult Behavior Rating Inventory of Executive Function (BRIEF-2A) will be used to measure these cognitive abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Solomon, PhD, MBA, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis MIND Institute, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. All collected data will be used solely for this study and will remain confidential in accordance with the IRB protocol.

REFERENCES:
- [Background] Drake RE, Bond GR, Goldman HH, Hogan MF, Karakus M. Individual Placement And Support Services Boost Employment For People With Serious Mental Illnesses, But Funding Is Lacking. Health Aff (Millwood). 2016 Jun 1;35(6):1098-105. doi: 10.1377/hlthaff.2016.0001. PMID 27269028
- [Background] Bond GR, Becker DR, Drake RE, Rapp CA, Meisler N, Lehman AF, Bell MD, Blyler CR. Implementing supported employment as an evidence-based practice. Psychiatr Serv. 2001 Mar;52(3):313-22. doi: 10.1176/appi.ps.52.3.313. PMID 11239097
- [Background] Bond GR, Drake RE, Becker DR. Generalizability of the Individual Placement and Support (IPS) model of supported employment outside the US. World Psychiatry. 2012 Feb;11(1):32-9. doi: 10.1016/j.wpsyc.2012.01.005. PMID 22295007
- [Background] Drake RE, Bond GR, Mascayano F. Modification of the Individual Placement and Support Model of Supported Employment. Psychiatr Serv. 2023 Jun 1;74(6):656-658. doi: 10.1176/appi.ps.20220484. Epub 2023 Jan 31. PMID 36718603
- [Derived] Solomon M, Yon-Hernandez JA, Ruder S, McGurk SR, Tancredi D, Takarae Y, Stahmer AC. A randomized controlled trial protocol for evaluating the feasibility, acceptability, and work outcomes of individualized placement and support adapted for autistic adults in the community. Contemp Clin Trials Commun. 2025 Aug 19;47:101536. doi: 10.1016/j.conctc.2025.101536. eCollection 2025 Oct. PMID 40893727